CLINICAL TRIAL: NCT00263484
Title: An International, Multicenter, Non-Randomized, Open-Labeled Study to Evaluate the Efficacy of Lower Dose Dexamethasone/Thalidomide and Higher Frequency ZOMETA(TM) in the Treatment of Previously Untreated Patients With Multiple Myeloma
Brief Title: Higher Frequency Zoledronic Acid in the Treatment of Multiple Myeloma
Acronym: dtZ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gleneagles Hospital (Other)
Collaborators: Singapore General Hospital (Other); National Cancer Centre, Singapore (Other); Tan Tock Seng Hospital (Other); Seoul National University Hospital (Other); Asan Medical Center (Other); Samsung Medical Center (Other); Chonnam National University Hospital (Other); Christian Medical College, Vellore, India (Other); Tata Memorial Hospital (Other Government)
Responsible Party: Dr Gerrard Teoh, Gleneagles Hospital, Singapore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SQMM01(dtZ)
Record Dates: First submitted 2005-12-07; First posted 2005-12-08 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Multiple Myeloma
Keywords: Steroids, Fluorinated; Thalidomide; Bisphosphonates
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Thalidomide; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- "dtZ" regimen, Initial therapy (Experimental): To test the efficacy of the "dtZ" regimen in previously untreated patients with multiple myeloma.
  Interventions: Drug: dexamethasone; Drug: thalidomide; Drug: zoledronic acid

INTERVENTIONS:
Drug: dexamethasone — 20 mg, PO (orally) on days 1-4, 8-11 and 15-18 of each 21 day cycle. 6 Cycles: until progression or unacceptable toxicity develops.
  Other Names: DEXAMETHASONE BEACONS
Drug: thalidomide — 100 mg, PO (orally) on days 1-21 of each 21 day cycle. 6 Cycles: until progression or unacceptable toxicity develops.
  Other Names: THALOMID (PHARMION); THADO (TTY)
Drug: zoledronic acid — 4 mg, IV (in the vein) on day 1 of each 21 day cycle. 6 Cycles: until progression or unacceptable toxicity develops.
  Other Names: ZOMETA

SUMMARY:
The purpose of this study is to determine whether lower than conventional doses of dexamethasone and thalidomide; and a higher dosing frequency of zoledronic acid are effective in the treatment of newly-diagnosed multiple myeloma.

DETAILED DESCRIPTION:
Patients with newly-diagnosed multiple myeloma (MM) may be treated using monthly cycles of dexamethasone plus thalidomide (DT). Unfortunately, the use of conventional doses of DT is associated with significant treatment-related morbidity and mortality, which is comparable to that observed with conventional chemotherapy. Hence, for safety reasons, patients frequently receive lower than conventional doses of DT (i.e. dt), and potentially experience a poorer anti-MM effect. The highly-potent aminobisphosphonate, zoledronic acid (Z), has been shown in pre-clinical mouse models to exhibit an impressive anti-MM effect. It is therefore possible to combined dt with Z (i.e. dtZ) to enhance the efficacy of (lower dose) dt. In addition, the anti-tumor effect of dtZ may potentially be augmented by using Z at a higher (three-weekly) dosing frequency.

ELIGIBILITY:
Inclusion Criteria:

* Age at or above 21 years
* Clinical diagnosis of MM
* Active MM with measurable disease
* Signed written informed consent
* Signed consent for drug safety program for thalidomide

Exclusion Criteria:

* Patients with Monoclonal Gammopathy of Undetermined Significance (MGUS)
* Patients with Indolent MM (IMM), or Smouldering MM (SMM)
* Known hypersensitivity (including severe cutaneous reactions) to d, t or Z
* Fulminant sepsis
* Females in the reproductive age group who refuse contraception
* Pregnancy
* 24 hr urinary creatinine clearance time (CCT) <30 ml/min
* Previous renal transplantation
* Severe peripheral neuropathy
* Recurrent DVT or PE
* Severe arrhythmias and cardiac conduction disorders
* Liver dysfunction of active viral hepatitis
* Osteonecrosis of the jaws (ONJ)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2005-12; Primary Completion 2008-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
1. To determine response rates (RR) and disease progression rates in all MM patients treated with dtZ regimen. | 4 months

SECONDARY OUTCOMES:
To assess overall survival (OS) in all patients treated with dtZ regimen. | 4 months
Assessment of incidence of skeletal related events (SREs). | 4 months
Assessment of percent change in renal function in all patients. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerrard Teoh, MD, Study Chair — Gleneagles Hospital, Singapore
Locations (10):
- India (2):
  - Tata Memorial Hospital, Mumbai, Mumbai
  - Christian Medical College, Vellore, Tamil Nadu
- Singapore (4):
  - Singapore General Hospital, Singapore
  - National Cancer Centre, Singapore, Singapore
  - Gleneagles Hospital, Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore, Singapore
- South Korea (4):
  - Chonnam National University Hwasun Hospital, Gwangju, Gwangju
  - Seoul National University Hospital, Seoul, Seoul
  - Samsung Medical Center, Seoul, South Korea, Seoul, Seoul
  - ASAN Medical Center, University of Ulsan, South Korea, Seoul, Seoul

REFERENCES:
- [Background] Yaccoby S, Pearse RN, Johnson CL, Barlogie B, Choi Y, Epstein J. Myeloma interacts with the bone marrow microenvironment to induce osteoclastogenesis and is dependent on osteoclast activity. Br J Haematol. 2002 Feb;116(2):278-90. doi: 10.1046/j.1365-2141.2002.03257.x. PMID 11841428
- [Background] Rosen LS, Gordon D, Kaminski M, Howell A, Belch A, Mackey J, Apffelstaedt J, Hussein MA, Coleman RE, Reitsma DJ, Chen BL, Seaman JJ. Long-term efficacy and safety of zoledronic acid compared with pamidronate disodium in the treatment of skeletal complications in patients with advanced multiple myeloma or breast carcinoma: a randomized, double-blind, multicenter, comparative trial. Cancer. 2003 Oct 15;98(8):1735-44. doi: 10.1002/cncr.11701. PMID 14534891
- [Background] Rajkumar SV, Hayman S, Gertz MA, Dispenzieri A, Lacy MQ, Greipp PR, Geyer S, Iturria N, Fonseca R, Lust JA, Kyle RA, Witzig TE. Combination therapy with thalidomide plus dexamethasone for newly diagnosed myeloma. J Clin Oncol. 2002 Nov 1;20(21):4319-23. doi: 10.1200/JCO.2002.02.116. PMID 12409330
- [Background] Weber D, Rankin K, Gavino M, Delasalle K, Alexanian R. Thalidomide alone or with dexamethasone for previously untreated multiple myeloma. J Clin Oncol. 2003 Jan 1;21(1):16-9. doi: 10.1200/JCO.2003.03.139. PMID 12506164
- See also: Clinic for Blood Disorders and Research (CBD), Gleneagles Hospital, Singapore — http://www.cbd.sg